CLINICAL TRIAL: NCT00821873
Title: Evaluation of the Composite of Cancellous and Demineralized Bone Plug (CR Plug) for Repair of Defects Created at the Harvest Site During the Osteochondral Autograft Transfer System(OATS)Procedure
Brief Title: Evaluation of the CR Plug for Repair of Defects Created at the Harvest Site From an Autograft in the Knee.
Acronym: CRB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRB2008; WIRB #20080290 (Other: Western IRB)
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Results first posted 2013-11-06 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Knee Injury
Keywords: Cartilage injury; OATS; Knee injury; allograft; autograft
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CR Plug BackFill (Experimental): Evaluation of the CR Plug for Repair of Defects Created at the Harvest Site
  Interventions: Other: CR Plug

INTERVENTIONS:
Other: CR Plug — CR Plug will be placed in the harvest site

SUMMARY:
The main objective of this study is to test the ability of an allograft plug to provide a successful repair of an osteochondral defect left at the harvest site during OATS procedure.

DETAILED DESCRIPTION:
The objective of this study is to determine how effective a plug made out of human bone (called "CR-Plug") will be in the treatment at the site that your tissue was removed, thereby filling the hole created during the OATS procedure.At the present, OATS is used for knee articular cartilage defects or injuries smaller than the size of a dime (or 2.5 cm2) in the areas that bear weight have been commonly treated by using a tiny cylinder of the subjects' own tissue called an osteochondral autograft (OATS).

ELIGIBILITY:
Inclusion Criteria:

* Are male or female at least 18 years of age and up to 55 years of age
* Must be skeletally mature
* Have a grade III or IV lesion in femoral condyle

Exclusion Criteria:

* Skeletally immature
* Osteoarthritic knees, osteonecrotic knees, osteophyte formation
* Use of any investigational therapy within thirty (30) days prior to the first visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2008-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Carter, MD, Principal Investigator — The Orthopedic Clinic, Assoc; David Flanigan, MD, Principal Investigator — The Ohio State Univesity; Phillip Stull, MD, Principal Investigator — Colorado Orthopedic Consultants; Jeffrey Dugas, MD, Principal Investigator — American Sports Medicine Institute
Locations (4):
- United States (4):
  - American Sports Medicine Institute, Birmingham, Alabama
  - The Orthopedic Clinic Assoc, Phoenix, Arizona
  - Colorado Orthopedic Consultants, Englewood, Colorado
  - Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from the patient population at the four investigative sites
Pre-assignment Details: This was a single arm study, thus there is no assignment
Period: Overall Study
Arm/Group | CR Plug BackFill
Started | 9
Completed | 5
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | CR Plug BackFill
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: MRI to Evaluate Success of Outcome.
Description: The CR-Plug to repair the harvest site defect left during the OATS procedure, the harvest site will be evaluated at 24 months post-operatively.
  The MRI scans were evaluated by a radiologist for several categories and these were then scored and transformed to an index, resulting in an outcome score ranging from 0-100 In this scale, 0 is the worst possible and 100 is the best possible score.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR Plug BackFill
Number analyzed (Participants) | 5
units on a scale | 88.6 (5.7)

ADVERSE EVENTS:
Groups:
- Adverse Events: Evaluation of the CR Plug for Repair of Defects Created at the Harvest Site
Arm/Group | Adverse Events
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=9)
Collapse of Graft (Musculoskeletal and connective tissue disorders) | 1 (1) — Interval Collapse in Size of Central Defect within the Anterior Lateral Femoral Condyle (per MRI)
PAIN IN RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1 (1) — NOT related
VOMITING NAUSEA (Gastrointestinal disorders) | 2 (2) — unlikely related
MEDICATION REACTION (General disorders) | 1 (1) — NOT related
DIARRHEA (Gastrointestinal disorders) | 2 (2) — NOT RELATED
FELL ON KNEE (Musculoskeletal and connective tissue disorders) | 1 (1) — NOT RELATED
PAIN RIGHT KNEE FROM FALL (Musculoskeletal and connective tissue disorders) | 1 (1) — NOT related
PAIN IN RIGHT KNEE FORM COLD (Musculoskeletal and connective tissue disorders) | 1 (1) — UNLIKELY RELATED
SWELLING IN RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1 (1) — NOT RELATED
ABDOMINAL PAIN (General disorders) | 1 (1) — NOT RELATED
TRANSIENT KNEE EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) — UNLIKELY RELATED
CHEST PAIN (General disorders) | 1 (1) — NOT RELATED
INFECTION OF LEFT KNEE (Musculoskeletal and connective tissue disorders) | 1 (1) — UNLIKELY RELATED
RIGHT LEG SWELLING (General disorders) | 1 (1) — NOT RELATED
INCREASED KNEE EFFUSION DUE TO FALL (Musculoskeletal and connective tissue disorders) | 1 (1) — NOT RELATED
DEPRESSION (Psychiatric disorders) | 1 (1) — NOT RELATED
QUADRICEPS ATROPHY - IPSILATERAL LEG (Musculoskeletal and connective tissue disorders) | 1 (1) — UNLIKELY RELATED
KIDNEY STONES (General disorders) | 1 (1) — NOT RELATED

LIMITATIONS AND CAVEATS:
Enrollment was closed early due for 2 factors:

1) Slow enrollment and 2) A potential change in the regulatory pathway for allografts used in cartilage repair.

Of the 9 patients enrolled, 4 were lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less